CLINICAL TRIAL: NCT00754858
Title: Phase II Study of Camtobell Inj.(Belotecan) in Combination With Cisplatin in Patients With Previously Untreated, Extensive-stage Small-cell Lung Cancer
Brief Title: Belotecan and Cisplatin in Treating Patients With Previously Untreated, Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000614308; YONSEI-4-2008-0127; CKDPC-YONSEI-4-2008-0127; YONSEI-07-YUHS-02
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — belotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- belotecan and Cisplatin (Experimental): belotecan 0.5 mg/m2 and Cisplatin 60mg/m2
  Interventions: Drug: belotecan hydrochloride; Drug: cisplatin

INTERVENTIONS:
Drug: belotecan hydrochloride
Drug: cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Belotecan may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving belotecan together with cisplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well belotecan works when given together with cisplatin in treating patients with previously untreated extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the antitumor efficacy, in terms of objective response rate, of belotecan hydrochloride and cisplatin in patients with previously untreated extensive-stage small cell lung cancer.

Secondary

* To assess additional evidence of antitumor activity as measured by overall and progression-free survival of these patients.
* To determine the safety and tolerability of this drug combination in these patients.

OUTLINE: Patients receive cisplatin IV on day 1 and belotecan hydrochloride IV on days 2-4.Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed small cell lung cancer meeting the following criteria:

  * Extensive-stage disease
  * Previously untreated disease
* At least one measurable disease
* No brain or leptomeningeal metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 mg/dL
* ALT and AST ≤ 2.0 times upper normal limit (ULN) (≤ 5.0 times ULN in the presence of liver metastasis)
* Alkaline phosphatase ≤ 2.0 times ULN
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* No active infection requiring intravenous antibiotics
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or in situ cancer
* No other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, interfere with the interpretation of study results, or make the patient ineligible for study entry, in the judgment of the investigator

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No other concurrent chemotherapy, radiotherapy, or immunotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Response rate as assessed by RECIST criteria | 21days(1cycle)
Overall survival | 21days(1cycle)
Progression-free survival | 21days(1cycle)
Hematologic and non-hematologic toxicity as assessed by NCI CTCAE v3.0 | 21days(1cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hang Kim, MD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea